CLINICAL TRIAL: NCT02636855
Title: A Screening Protocol to Determine Tumor Antigen Expression and HLA Sub-Type for Eligibility Determination for Clinical Trials Evaluating the Safety and Efficacy of Autologous T Cells Expressing Enhanced TCRs in Subjects With Solid and Hematological Malignancies
Brief Title: Screening Protocol for Tumor Antigen Expression Profiling and HLA Typing for Eligibility Determination
Status: Completed | Type: Observational
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Other Study IDs: ADP-0000-001
Record Dates: First submitted 2015-11-23; First posted 2015-12-22 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Solid and Hematological Malignancies
Keywords: Solid and Hematological Malignancies; Screening; Metastatic; Previously Treated; MAGE-A4; Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
This screening study is intended for men and women ≥ 18 to ≤ 75 years of age who have advanced solid or hematologic malignancy. The study will assess a subject's human leukocyte antigen (HLA) subtype and tumor antigen expression profile. Based on the results, it will be determined if a subject is eligible to be considered for Adaptimmune sponsored clinical trials testing the safety and efficacy of genetically changed T cells targeting specific tumor antigens. No treatment intervention will occur as part of this screening study.

Upon enrollment, subjects will be required to provide a blood sample for HLA subtype analysis. If the results of the analysis match the HLA-A subtypes noted in the inclusion criteria and do not express the HLA subtypes that are exclusionary for the available interventional clinical trial(s), then the subject will be required to provide either an archival tumor specimen or fresh tumor tissue biopsy. The tumor specimen will be screened at a central laboratory for the expression (protein or gene) of multiple antigens which may include, but are not limited to MAGE-A4. Based upon the results of these diagnostic analyses, if eligible, subjects will be referred to an appropriate available interventional clinical trial(s) at the discretion of the Investigator.

Following screening, tumor samples will be retained by Adaptimmune for the purpose of developing and validating in vitro diagnostic (IVD) assay(s) for antigen expression profiling which is required for regulatory approval of a new therapeutic product indication.

DETAILED DESCRIPTION:
This multicenter screening study will be conducted in order to determine a subject's tumor antigen expression profile and HLA subtype, and subsequent eligibility for Adaptimmune sponsored clinical treatment trials studying the safety and efficacy of autologous genetically modified T-cells engineered with enhanced TCRs targeting specific antigens. No treatment intervention will occur as part of this screening study. Specific Adaptimmune sponsored interventional protocols have been designated to utilize this screening protocol to determine preliminary eligibility. Therefore, details of the available interventional clinical trial(s) (e.g., HLA subtype, tumor antigen, and other eligibility criteria) should be understood before consenting subjects for this screening protocol.

For this screening study, subjects with confirmed advanced solid or hematologic malignancy or recurrent disease, as described in the respective Adaptimmune clinical trial protocol(s), will be required to provide a blood sample for diagnostic analysis. The blood sample will be used for HLA subtype analysis. If the results of the analysis match the HLA subtype specified in the available interventional clinical trial(s), then the subject will be required to provide either an archival tumor specimen or fresh tumor tissue biopsy. The tumor specimen will be screened at a central laboratory for the expression (gene or protein) of multiple antigens using Clinical Trial Assays. The Clinical Trial Assays to be used in this protocol have undergone CLIA validation to establish the sensitivity, specificity and performance of the assays. The antigens to be screened may include, but are not limited to the following: NY-ESO-1 and/or LAGE-1a and MAGE-A10. Based upon both the tumor antigen expression and the HLA subtype, if eligible, subjects will be referred to appropriate available interventional trial(s) at the discretion of the Investigator.

The secondary objective of the study is the collection and analysis of tumor tissue specimens to enable the development and validation of single and/or multiple-marker ('multiplex') IVD assay(s) for antigen expression profiling. It is a regulatory requirement to develop the IVD(s) as a companion diagnostic(s) to accompany a future new indication drug application(s). Therefore all tumor specimens from this study will be retained by Adaptimmune for companion diagnostic validation purposes.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent;
2. Histologically or cytologically confirmed diagnosis of advanced solid or hematologic malignancy or recurrent disease, as described in the respective Adaptimmune clinical treatment protocol (including, but not limited to myeloma, melanoma, NSCLC, head and neck, gastric and bladder cancer);
3. Male or female ≥ 18 to ≤75 years of age;
4. Life expectancy > 3 months;
5. Ability to provide a blood sample;
6. Ability to provide one of the following tumor tissue samples:

   i. formalin-fixed, paraffin-embedded (FFPE) tumor block or tissue sections from a current lesion/the most current setting, OR

ii. a fresh biopsy is feasible, OR;

iii. a FFPE archival primary tumor block or tissue sections

Exclusion Criteria:

1. Any bleeding diathesis or coagulopathy, which at the discretion of the Investigator may put the subject at risk.
2. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the screening study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with confirmed diagnosis of advanced solid or hematologic malignancy or recurrent disease
Sampling Method: Non-Probability Sample
Enrollment: 9122 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with the expression (gene or protein) of multiple antigens (including, but are not limited to MAGE-A4 , and others) [ Time Frame: 10 years ] | 10 years
  To screen subject tumor tissue in order to determine their tumor antigen expression profile, and HLA subtype, for subsequent assessment of eligibility for various Adaptimmune sponsored targeted T cell therapy clinical trials.

SECONDARY OUTCOMES:
Retention of screening tumor tissue for the future development and validation of single and/or multi-plex companion diagnostic platforms for the detection of tumor antigen expression. [ Time Frame: 10 years ] | 10 years
  Following screening for the antigen expression profile, remaining screening tissue will be used for the purpose of developing and validating companion diagnostic assays for antigen screening for regulatory approval. Tumor tissue will be used for the analytical validation (which includes testing for efficiency, sensitivity, specificity, exclusivity, accuracy and precision), as well as the clinical validation of such diagnostic assays.

OTHER OUTCOMES:
Incidence of antigen expression in solid and hematological malignancies [ Time Frame: 10 years ] | 10 years
  To collect data regarding the frequency of occurrence of antigens in tumor tissue samples of different tumor types.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (25):
  - City of Hope, Duarte, California
  - Stanford Cancer Institute (Stanford University), Stanford, California
  - Boca Raton Regional Hospital, Lynn Cancer Institute, 701 NW 13th Street, Boca Raton, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Patricia D. and M. Scot Kaufman Cancer Center, Bel Air, Maryland
  - UMD St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Duke Cancer Institute, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology- Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (8):
  - University Hospital of Navarra (Pamplona), Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario 12 Octubre Avda. de Córdoba s/n, Madrid
  - Centro Integral Oncológico Clara Campal, HM CIOCC (START MADRID-CIOCC), Madrid
  - Hospital Virgen del Rocio, Sevillia, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - University College Hospital Macmillan Cancer Centre, London
  - The Christie NHS Foundation Trust, Manchester